CLINICAL TRIAL: NCT03718455
Title: Evaluation of Magseed as Localization Device for Biopsy Proven Metastatic Axillary Lymph Nodes in Women With Breast Cancer
Brief Title: Evaluation of Magseed as Localization Device for Biopsy Proven Metastatic Axillary Lymph Nodes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Limited operating room availability
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Genevieve A. Woodard, Senior Associate Consultant, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18-004803
Record Dates: First submitted 2018-10-15; First posted 2018-10-24 (Actual); Results first posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Single cohort of twenty women receiving neoadjuvant chemotherapy with breast cancer will have a Magseed inserted into a biopsy proven metastatic axillary lymph node for pre-surgical localization. The Magseed is a FDA approved device for pre-surgical localization and has been recently approved for use in the axilla and for placement longer than 30 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Axillary Magseed (Experimental): Single cohort of twenty women receiving neoadjuvant chemotherapy with breast cancer will have a Magseed inserted into a biopsy proven metastatic axillary lymph node for pre-surgical localization.
  Interventions: Device: Axillary Magseed

INTERVENTIONS:
Device: Axillary Magseed — The Magseed will replace the investigators' current clinical practice of using radioactive seeds in women receiving neoadjuvant chemotherapy.

SUMMARY:
Currently, breast cancer patients who are treated with neoadjuvant chemotherapy (NAC) before surgery may have a biopsy clip placed in the lymph node at the time of or shortly after percutaneous biopsy. Following 12-20+ weeks of NAC, pre-surgical localization of the sampled axillary lymph node using a radioactive seed can be done up to 5 days prior to surgery. Localization of the sampled lymph node in patients with complete imaging response to NAC can be technically challenging if the biopsy clip is not sonographically visible. This study is designed to see if it is feasible to place a Magseed, which is magnetic seed, into the abnormal node either at the time of fine needle aspiration (FNA) or after NAC, just prior to surgery, and to be able to accurately identify the abnormal node at the time of surgery.

DETAILED DESCRIPTION:
Part 1: Ten women with biopsy proven breast cancer and metastasis to an axillary lymph node will have a Magseed placed into the metastatic lymph node AFTER neoadjuvant chemotherapy (NAC) and just prior to surgery. These patients will have a non-contrast enhanced breast MRI development study to evaluate and identify ways to reduce the artifact in the axilla created by the Magseed. Efficacy of the localization with the Magseed will be available within a week of the placement.

Part 2: Ten additional women with biopsy proven breast cancer and metastasis to an axillary lymph node will have a Magseed placed into the metastatic lymph node BEFORE NAC. These patients will have routine contrast enhanced MRIs, mammograms, and ultrasounds before and after NAC to evaluate treatment response.

Seed placement: Once a patient has been identified eligible for the research study and has provided written informed consent the patient will have a Magseed placed into the biopsy proven lymph node. The Magseed delivery system is identical to the investigators' current practice using radioactive seeds. The seed is pre-loaded into the needle and is inserted into the lymph node following local anesthesia with 1% lidocaine. Once the seed is deployed, post procedure seed location is confirmed sonographically and mammographically with tomosynthesis.

MRI: Ten no-charge limited non-contrast breast MRIs for research development purposes are available for this study through the radiology department. Phase 1 participants will enroll in the study after their pre- and post-NAC imaging has already been performed per routine clinical practice. These participants will have a single non-contrast enhanced breast MRI using the investigators' standard non-contrast sequences (axial ideal T1 and T2-weighted, axial Short-TI Inversion Recovery (STIR), and axial 3D vibrant using a dedicated breast coil, FOV 28 cm or to fit the patient size, and an image-thickness/image-increment of 5mm/1mm). A physicist will participate in the scanning of these patients to evaluate the extent of artifact in the axilla and adjacent breast tissue and optimize scanning parameters to reduce this artifact.

Phase 2 participants will enroll in the study prior to NAC and have routine contrast enhanced breast MRIs performed before and after NAC. Clinically indicated MRI scans will be charged to the patient's insurance company as this imaging is standard clinical practice. The MRI protocol will use the investigators' standard clinical sequences (axial ideal T1 and T2-weighted, axial STIR, and axial 3D vibrant using a dedicated breast coil). Once contrast is injected (gadobutrol 10mmol/10mL) 3D vibrant sequences will be obtained four times after contrast injection (FOV 28 cm or to fit the patient size, and an image-thickness/image-increment of 5mm/1mm).

Mammogram: Patients enrolled in the research study will have standard mammographic imaging before and after NAC, which will include both the breast and axilla as per routine clinical protocol.

Ultrasound: Patients enrolled in the research study will have standard sonographic imaging before and after NAC of the breast and axilla as per routine clinical protocol. Post-NAC ultrasound of the axilla will be a supplemental assessment to breast MRI as the Magseed artifact may obscure these findings.

Seed Removal: As per the current practice, patients will have targeted axillary lymph node dissection including both the localized lymph node and sentinel lymph node. Identifying the lymph node containing the Magseed will require the Sentimag handheld probe in the operating room. This device which functions similar to the gamma probe has been approved for an equipment trial starting in August of 2018. Once the lymph node has been excised a specimen radiograph will be obtained to verify removal.

ELIGIBILITY:
Inclusion Criteria:

1. Women 18 years or older
2. Neoadjuvant chemotherapy planned prior to surgical excision
3. Scheduled for target axillary lymph node dissection including the localized lymph node and sentinel lymph node

Exclusion Criteria:

1. Pregnant or nursing women
2. Allergy to lidocaine or gadolinium
3. Contraindication to MRI (i.e. pacemaker)
4. Axillary Infection
5. Prior axillary radiation
6. Known allergy to bone wax, beeswax or propolis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Genevieve A Woodard, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Axillary Magseed
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Axillary Magseed
Number analyzed (Participants) | 1
Age, Customized [Number; unit: participants]
  60 years old | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Evaluate if Magseed is a Viable Alternative to Radioactive Seed as a Localization Method for Biopsy Proven Metastatic Breast Carcinoma Following Neoadjuvant Chemotherapy.
Description: The rate of successful placement of the Magseed into the axilla in the radiology department will be measured. Any substantial barriers to placement compared to the investigators' current clinical practice with the radioactive seed will be subjectively gathered from the radiologist and will be reported on a case-by-case basis.
Time Frame: 2-22 weeks after placement of the Magseed
Population: Terminated study due to Limited operating room availability. Data was not analyzed
Arm/Group | Axillary Magseed
Number analyzed (Participants) | 0

2. Primary Outcome: Assess the Success of Retrieval of the Magseed and Biopsy Proven Metastatic Lymph Node in the Operating Room Compared to the Current Practice With the Radioactive Seed.
Description: The rate of successful retrieval of the Magseed from the axilla in the operating room will be measured. Any substantial barriers to retrieval compared to the investigators' current clinical practice with the radioactive seed will be subjectively gathered from the surgeon and will be reported on a case-by-cases basis.
Time Frame: 2-22 weeks after placement of the Magseed
Population: Terminated study due to Limited operating room availability. Data was not analyzed
Arm/Group | Axillary Magseed
Number analyzed (Participants) | 0

3. Secondary Outcome: Determine the Amount of Artifact Created by the Magseed in the Axilla at MRI and Identify Imaging Optimization to Minimize the Artifact Produced by the Magnetic Clip.
Description: The maximum dimension of the susceptibility artifact will be measured in centimeters with the investigator's current clinical MRI protocols. Additional MRI sequences with susceptibility artifact suppression techniques will be conducted and the maximum dimension of the susceptibility artifact will be measured in centimeters. Differences in these measurements will be analyzed.
Time Frame: 2-22 weeks after placement of the Magseed
Population: Terminated study due to Limited operating room availability. Data was not analyzed
Arm/Group | Axillary Magseed
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline to end of study, approximately two years for the subject.
Arm/Group | Axillary Magseed
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
Terminated study due to Limited operating room availability. Data was not analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-04): https://cdn.clinicaltrials.gov/large-docs/55/NCT03718455/Prot_SAP_000.pdf